CLINICAL TRIAL: NCT00472953
Title: Inhaled Pre-prandial Human Insulin Versus Subcutaneous Injected Insulin Aspart in Subjects With Diabetes and Chronic Obstructive Pulmonary Disease: A 52-week Open Label, Multicentre, Randomized, Parallel Trial to Investigate Long-term Safety
Brief Title: Safety of Inhaled Human Insulin in Subjects With Diabetes Mellitus and Chronic Obstructive Pulmonary Disease (COPD)
Acronym: iINHALE 8
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1617; 2006-004731-29 (EudraCT Number)
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: inhaled human insulin
- B (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: inhaled human insulin — Treat-to-target dose titration scheme, pre-prandial, inhalation.
  Arms: A
Drug: insulin aspart — Treat-to-target dose titration scheme, pre-prandial, injection s.c.
  Arms: B

SUMMARY:
This trial is conducted in Europe, Asia and South America. A one-year clinical trial to compare the safety of inhaled human insulin to subcutaneous insulin aspart in subjects with type 1 or type 2 diabetes and chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease
* Type 1 or type 2 diabetes
* HbA1c lower or equal to 11.0 %
* Body Mass Index (BMI) lower or equal to 40.0 kg/m2

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Current smoking or smoking within the last 6 months
* Other pulmonary disease including asthma
* Proliferative retinopathy or maculopathy requiring acute treatment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-05-15 (Actual); Primary Completion 2008-03-05 (Actual); Study Completion 2008-03-05 (Actual)

PRIMARY OUTCOMES:
To evaluate pulmonary safety comparing inhaled insulin to subcutaneous injections | After one year

SECONDARY OUTCOMES:
Patient Reported Outcomes | After one year
Diabetes control measured by change in HbA1c from baseline | After one year
Preprandial Insulin Doses | After one year

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (21):
- Argentina (2):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Ciudad de Buenos Aires
- India (6):
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Mumbai
  - Novo Nordisk Investigational Site, Pune
- Novo Nordisk Investigational Site, Bucharest, Romania
- Slovakia (4):
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Ľubochňa
  - Novo Nordisk Investigational Site, Moldava nad Bodvou
  - Novo Nordisk Investigational Site, Žilina
- Taiwan (3):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Chiayi City
  - Novo Nordisk Investigational Site, Taipei
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Erzurum
  - Novo Nordisk Investigational Site, Gaziantep
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Kocaeli

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com